CLINICAL TRIAL: NCT06279260
Title: National Robotics-Assisted Radical Prostatectomy Database: Exploring Learning Curves and Long Term Surgical, Oncological and Patient Reported Outcome Measures (PROMS)
Brief Title: National Robotics-Assisted Radical Prostatectomy Database
Acronym: RASOR
Status: Recruiting | Type: Observational
Sponsor: Melbourne Health (Other)
Collaborators: Peter MacCallum Cancer Centre, Australia (Other); Epworth Healthcare (Other); St Vincent's Hospital (Other); Austin Health (Other Government); Barwon Health (Other Government); Ballarat Health Services (Other); Western Health, Australia (Other Government)
Responsible Party: Principal Investigator, Nathan Lawrentschuk, Professor, Melbourne Health
Other Study IDs: 104451/2023.295
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Database; Prostate Cancer; Robotic-assisted Radical Prostatectomy; Surgical Outcomes; Oncological Outcomes; Patient Reported Outcome Measures; Learning Curve
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In Australia, nearly 70 men are diagnosed with Prostate cancer every day. Prostate removal (Radical Prostatectomy) is the proven treatment option to control cancer spread. Most of the prostate removal surgeries are done using robots. Robotic assisted prostate removal surgeries have been invented to minimise the risk of side effects post-surgery. Doctors prefer the robots over open surgery as there are benefits to patients (shorter hospital stays, lesser blood loss and better quality of life) and surgeons (better dexterity, improved field of vision and less pain). However, the cost of the robot outweighs the benefits at present and there is very less information concerning the long-term outcomes for patients.

Studies conducted so far are small scale studies and the results from these studies cannot be generalized to the population at large in Australia. So, there is need for a largescale study that will look at the long-term outcomes and the factors that impact robotic surgeries across the metropolitan and rural hospital sectors.

Hence, this comprehensive database has been setup to collaborate with major hospitals, across metropolitan and rural areas in Australia. Through this database, researchers will be able to explore the diagnostic pathway for Prostate cancer and understand the long-term benefits of robotic surgery through patient reported questionnaires. Outcomes from this database will also help compare the quality of care against other powerhouses of robotic surgery.

Eventually, the database aims to standardize diagnostic pathways and clinical notes that are the same across different hospitals conducting robotic-assisted surgeries for Prostatectomy and improve care for prostate cancer patients across the country.

DETAILED DESCRIPTION:
Radical Prostatectomy (RP) is the only surgical option for resectable PCA with evidenced benefit for overall survival [5,6]. Robotic-Assisted Radical Prostatectomy (RARP) is an evolved RP represents a significant advancement in PCa treatment offering better field of vision & dexterity for the surgeons [7,8,9,10,11] compared to other procedures such as Open Radical Prostatectomy (ORP) and Laparoscopic Radical prostatectomy (LRP).

A meta-analysis [12] of Randomized Control Trials (RCT) and non-randomized studies reported that RARP and LRP were similar in terms of blood loss, catheter indwelling time, overall complication rate, overall positive surgical margin and biochemical recurrence rates. However, quantitative synthesis of non-randomized studies indicated that RARP was associated with better functional and oncological outcomes compared to LRP.

Despite RARP holding promising benefits, it also presents some potential challenges such as:

1. Learning curve - Surgeons require significant training and experience to become proficient in using robotic systems. This learning curve can impact surgical outcomes, especially in less experienced hands.
2. Cost - The robotic systems and associated instruments are expensive, leading to higher upfront costs for hospitals. This can translate to higher costs for patients and healthcare systems.
3. Disparity between private and public sectors: availability of robotic surgery can be limited by geographic and economic factors, potentially leading to disparities in access to advanced surgical option.

A retrospective audit of all RARP procedures performed at high volume centre in Australia highlighted, operating time costs for RARP is $134.16 AUD per minute which costs the patient and the hospital $30, 588.48 AUD per case. The health industry average costs for a RARP procedure is 32,199 AUD per case. A transition point of 65 cases at the industry average will cost up to $2,092,935 AUD to consistent primary outcomes for patients [13]. Surgeon's experience and efficiency become an important determinant of post RARP outcomes. Incorporating assessment protocols and intensive training programs might contribute to better post RARP outcomes [14].

Another Australian study [15] evaluated the ORP versus RARP outcomes at a high-volume centre. Results of the study indicated significantly lower mean Length of Stay (LOS) for RARP compared with ORP (1.2 vs 4.4 days) and a much higher readmission rate after ORP (19%) compared with RARP (2%). Though the study reported evidenced benefits, it also highlighted that case-mix funding model failed to adequately reimburse the public hospitals for RARP when compared with ORP despite efficient use of hospital resources in terms of hospital stay and reduction in costly readmissions.

A massive inequality gap exists between the public and private sectors. A retrospective analysis of Victorian Cancer Registry data found proportion of private patients who underwent radical prostatectomy (44%) was larger than that for public patients (28%). [16] There are fewer robots in the public sector compared to private hospitals hence public patients are offered alternate approaches.

A barrier to the uptake of robotic-assisted surgery (RAS) continues to be the perceived high costs. A lack of detailed costing information has made it difficult for public hospitals in particular to determine whether use of the technology is justified [17]. This inconsistency in approach and lack of detail makes it difficult for local hospital administrators, health ministries and governing bodies to determine whether the costs of the technology are reasonable and worth the ongoing investment, and has the potential to impact on future strategic decision-making.

It is notable, that robust evidence substantiating the advantages of robotic surgery from high volume centres is currently insufficient. The acquisition of high-quality evidence pertaining to surgical techniques poses a formidable challenge [18]. Robust investigations, characterized by substantial scale and comparativeness, are imperative for a comprehensive assessment of the surgical, oncological and Patient reported outcomes along with learning curves of surgeons associated with RARP.

There is an imperative need for the establishment of a population-based database that systematically captures a comprehensive array of surgical operatives, learning curves of surgeons and the patient-reported quality of life measures (PROM). A structured database holds the potential to provide a standardized framework, enabling robust comparative analyses, trend identification, and the formulation of evidence-based guidelines for the individualized management of prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this database, an individual must meet all of the following criteria:

1. Individuals who consent to participate,
2. within the age range of 18 to 90 years,
3. confirmed diagnosis of localized prostate cancer (PCa)
4. patients receiving medical attention at hospitals engaged in collaborative efforts with the designated database.

Exclusion Criteria:

1. Participants are not eligible to take part in the database:
2. Individuals who have not undergone robotic surgery for prostatectomy or TP biopsy. ,
3. without a diagnosis of prostate cancer or
4. who decline to provide consent for the collection of their health information
5. Under the age of 18 years.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males who are diagnosed with localized Prostate cancer
Study Population: The database will entail recruitment of retrospective and prospective patient cohorts to collect and analyse data. Retrospective data from the last five years will be obtained from the medical records. Prospective data will be collected from each participating site.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2050-12 (Estimated); Study Completion 2050-12 (Estimated)

PRIMARY OUTCOMES:
To provide a standardized framework, enabling robust evidence strengthening & analyses, trend identification, and the formulation of evidence-based guidelines for the individualized management of PCa. | At baseline, 4 weeks, 6 months, 12 months, 24 months and 36 months post-surgery.
  Standardize notes that are the same across different hospitals conducting robotic-assisted surgeries for prostatectomy.

SECONDARY OUTCOMES:
Patient reported quality of life outcome measures | At baseline, 4 weeks, 6 months, 12 months, 24 months and 36 months post-surgery.
  The first set of outcome variables will be the functional outcomes from the PROMs, using the Expanded Prostate Cancer Index Composite (EPIC)-26 questionnaire
Surgical | At baseline, 4 weeks, 6 months, 12 months, 24 months and 36 months post-surgery.
  The second set of outcome variables will gather detailed insights into surgical measures in In terms of operative and post-operative characteristics.
Oncological | 4 weeks, 6 months, 12 months, 24 months and 36 months post-surgery.
  The third set of outcome variables will collect the oncological measures in terms of Biochemical re-occurrence and margin status.

CONTACTS AND LOCATIONS:
Locations (8):
- Australia (8):
  - Ballarat Health, Ballarat, Victoria
  - Barwon health, Geelong, Victoria
  - Austin Healthcare, Melbourne, Victoria
  - E.J Whitten Prostate Cancer Centre, Epworth Healthcare, Melbourne, Victoria
  - St. Vincent's Private Hospital, Melbourne, Victoria
  - Western Heath, Melbourne, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No
* Patient data will only be transferred and analysed in a coded form by mentioned investigators.
  * Transferring patient data will require host organisation's formal approval
  * Individual patients will not be identifiable from the presented or published material.
  * The institution and the researcher must comply with all relevant laws and standards in relation to the use of the material.
  * The institution and researcher must not use the material for any purpose other than the specified research or other purposes expressly permitted under the terms of the Agreement.
  * Data linkage across sites will be set up when necessary. Once linkage has been completed, identifiers will be removed from the data to be used in the research, unless consent has been given for its identifiable use.

REFERENCES:
- [Background] Perera S, Fernando N, O'Brien J, Murphy D, Lawrentschuk N. Robotic-assisted radical prostatectomy: learning curves and outcomes from an Australian perspective. Prostate Int. 2023 Mar;11(1):51-57. doi: 10.1016/j.prnil.2022.10.002. Epub 2022 Oct 29. PMID 36910896
- [Background] Fridriksson JO, Folkvaljon Y, Lundstrom KJ, Robinson D, Carlsson S, Stattin P. Long-term adverse effects after retropubic and robot-assisted radical prostatectomy. Nationwide, population-based study. J Surg Oncol. 2017 Sep;116(4):500-506. doi: 10.1002/jso.24687. Epub 2017 Jun 7. PMID 28591934
- [Background] Tiruye T, O'Callaghan M, Moretti K, Jay A, Higgs B, Santoro K, Boyle T, Ettridge K, Beckmann K. Patient-reported functional outcome measures and treatment choice for prostate cancer. BMC Urol. 2022 Nov 5;22(1):169. doi: 10.1186/s12894-022-01117-1. PMID 36335325
- [Background] Chandrasekar T, Tilki D. Prostate cancer: Comparing quality of life outcomes after prostate cancer treatment. Nat Rev Urol. 2017 Jul;14(7):396-397. doi: 10.1038/nrurol.2017.81. Epub 2017 Jun 13. No abstract available. PMID 28607497